CLINICAL TRIAL: NCT05790460
Title: Telehealth Based Synchronous Navigation to Improve Molecularly-Informed Care for Patients With Lung Cancer
Acronym: TESTING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Charu Aggarwal, Associate Professor of Medicine, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPCC 22522; P50CA271338 (NIH); 852857 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2023-02-20; First posted 2023-03-30 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Molecular Testing; Lung Cancer; Telehealth; Liquid Biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Experimental): Patients in the intervention arm will be scheduled for an enhanced synchronous telehealth visit with a trained lung cancer nurse navigator prior to tissue biopsy. The enhanced synchronous telehealth visit will ideally occur between the initial clinical appointment and diagnostic biopsy (typically a period between two and seven days). In addition to the activities conducted as part of usual care, the nurse navigator will: 1) provide more detailed and individualized education on lung cancer and the rationale for comprehensive molecular testing, including plasma-based tests; and 2) if the patient agrees to testing, pend a default order for plasma-based molecular testing (if not already ordered) for the clinician to sign and arrange for phlebotomy to be performed at the time of the patient's tissue biopsy.
  Interventions: Other: Telehealth
- Usual Care (No Intervention): Patients in the usual care arm will receive a telephone call from a trained lung cancer nurse navigator after biopsy, as is typical at Penn Medicine, to 1) review the roles of clinicians on the medical oncology care team; 2) provide brief education on lung cancer; and 3) review the patient's diagnostic history and coordinate collection or completion of imaging required for guideline-recommended cancer staging. At the initial in-person oncology visit, the oncologist may choose to order plasma-based testing if appropriate (and if not already ordered or pending).

INTERVENTIONS:
Other: Telehealth — Enhanced synchronous telehealth nurse navigation, compared to usual care nurse navigation, to increase timely molecularly-informed treatment recommendations through early integration of concurrent molecular testing.
  Arms: Telehealth

SUMMARY:
The goal of this trial is to design and test a telehealth nurse navigation intervention for patients with suspected locally advanced/metastatic NSCLC to improve timely molecularly-informed treatment recommendations through early integration of concurrent molecular testing.

DETAILED DESCRIPTION:
The overarching goal of this pilot trial is to design and test a nurse navigation intervention delivered via telehealth for patients with suspected locally advanced/metastatic NSCLC to improve timely molecularly-informed treatment recommendations through early integration of concurrent molecular testing (i.e., tumor tissue and plasma-based molecular testing or plasma only when tumor tissue is insufficient/unavailable). The central hypothesis is that providing telehealth nurse navigation to support completion of concurrent molecular testing will result in higher rates of comprehensive testing, improved timeliness of molecularly-informed treatment recommendations (primary endpoint), earlier initiation of molecularly-informed treatment, more meaningful patient-clinician communication, and higher levels of overall satisfaction among patients and clinicians. Drawing from systematic evidence on the role of navigation for coordination of cancer care and informed by insights from communication science and behavioral economics, the specific telehealth strategy to be tested is synchronous telehealth nurse navigation in combination with default ordering of plasma-based testing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Based on cross-sectional imaging, suspected to have locally advanced/metastatic NSCLC (as determined by the evaluating clinician)
* Scheduled for an appointment in the lung cancer evaluation clinic

Exclusion Criteria:

* Are not suspected to have locally advanced/metastatic NSCLC
* Have a concurrent active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Charu Aggarwal, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment/randomization occurred from May 8, 2023 to November 8, 2023. On November 8, 2023, the study was paused and later terminated.
Period: Overall Study
Arm/Group | Telehealth | Usual Care
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telehealth | Usual Care | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [62 to 77] | 70 [64 to 78] | 68 [62 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 13 | 15 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 25 | 53
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 16 | 20 | 36
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Molecularly-informed Treatment Recommendations
Description: Receipt of a molecularly-informed treatment recommendation for patients with metastatic NSq NSCLC at the time of the patient's initial oncology visit.
Time Frame: Measured up to 12 weeks from randomization
Population: All participants who 1) were diagnosed with Stage IIIB/C (with palliative intent treatment) or Stage IV non-squamous NSCLC and 2) had an initial outpatient oncology evaluation within 12 weeks of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 5 | 6
Participants | 2 | 2

2. Secondary Outcome: Rate of Telehealth Visit Completion
Description: Telehealth visit completion defined as successful completion of a telehealth visit prior to biopsy
Time Frame: Measured up to 3 weeks from randomization
Population: All participants randomized to telehealth who underwent biopsy. One participant was excluded from this analysis due to not having a biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth
Number analyzed (Participants) | 27
Participants | 25

3. Secondary Outcome: Rate of Completion of Comprehensive Molecular Testing (Tissue and/or Plasma Testing) Prior to Initiation of First Line Therapy
Description: Rate of completion of comprehensive molecular testing (tissue and/or plasma testing) prior to initiation of first line therapy
Time Frame: Measured up to 12 weeks from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 28 | 27
Participants | 26 | 12

4. Secondary Outcome: Identification of One or More Targetable Mutations
Description: Identification of one or more targetable mutations
Time Frame: Measured up to 12 weeks from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 28 | 27
Participants | 2 | 2

5. Secondary Outcome: Timeliness of Molecularly-informed Treatment Recommendation
Description: Time from randomization to recommendation of a molecularly-informed treatment, as documented in the EMR
Time Frame: Measured up to 12 weeks from randomization
Population: Participants who received a molecularly-informed treatment recommendation up to 12 weeks from randomization.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 5 | 6
days | 17.6 [16 to 18] | 38.5 [27.5 to 43]

6. Secondary Outcome: Overall Survival
Description: Overall survival
Time Frame: Measured up to 1 year from the time of randomization to death from any cause
Population: All participants who 1) were diagnosed with Stage IIIB/C (with palliative intent treatment) or Stage IV non-squamous NSCLC and 2) chose active treatment, rather than hospice care, after diagnosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 6 | 6
Participants
  Alive | 5 | 4
  Deceased | 1 | 2

7. Secondary Outcome: Proportion of Patients With Diagnosis Other Than Metastatic Nonsquamous NSCLC (Telehealth Arm Only)
Description: Proportion of patients with diagnosis other than metastatic nonsquamous NSCLC (Telehealth arm only)
Time Frame: Measured at 12 weeks from randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth
Number analyzed (Participants) | 27
Participants | 21

8. Secondary Outcome: Time From Randomization to Treatment Initiation
Description: Time from randomization to treatment initiation
Time Frame: Measured at 12 weeks from randomization
Population: All participants who had active treatment initiation (excludes hospice) within 12 weeks of randomization.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 5 | 6
days | 27.6 [23 to 35] | 50.3 [38 to 67]

ADVERSE EVENTS:
Time Frame: 1 year from randomization
Arm/Group | Telehealth | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/6 | 3/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

LIMITATIONS AND CAVEATS:
Early termination due to insufficient accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT05790460/Prot_SAP_000.pdf